CLINICAL TRIAL: NCT06630845
Title: Comparison of Whole Body DWI to FDG PET Using PET/MRI
Brief Title: Comparison of Whole Body DWI to FDG PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Society of Abdominal Radiology (Other); GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24926; NCI-2024-09278 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Cancer
Keywords: Imaging Study
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Whole Body DWI plus FDG PET/MRI (Experimental): Participants will receive 5 to 10 Megabecquerel (MBq) +/- 10% of 18F-fluorodeoxyglucose as an intravenous injection and undergo a FDG PET/MRI scan that will extend from the vertex to the mid-thighs. Imaging will be performed from vertex to mid-thighs using standard protocol. Participants may also obtain an optional second FDG PET/MRI with DWI within 6 months.
  Interventions: Drug: Fluorodeoxyglucose F18; Procedure: Positron Emission Tomography combined with Magnetic resonance imaging (PET/MRI); Procedure: Whole Body Magnetic Resonance Imaging with Diffusion-Weighted Imaging (WB-MRI-DWI); Device: General Electric (GE) SIGNA PET/MR

INTERVENTIONS:
Drug: Fluorodeoxyglucose F18 — Given IV as part of routine imaging
  Other Names: Fludeoxyglucose F18 (FDG); 2-deoxy-2-[fluorine-18]fluoro-D-glucose; Fluorodeoxyglucose
Procedure: Positron Emission Tomography combined with Magnetic resonance imaging (PET/MRI) — Imaging procedure
  Other Names: PET/MRI
Procedure: Whole Body Magnetic Resonance Imaging with Diffusion-Weighted Imaging (WB-MRI-DWI) — Imaging procedure done concurrently with PET/MRI
  Other Names: WB-MRI-DWI
Device: General Electric (GE) SIGNA PET/MR — Imaging device
  Other Names: GE SIGNA PET/MR; SIGNA PET/MR

SUMMARY:
This is a single arm prospective trial that evaluates whole body diffusion weight imaging (DWI) compared to 18F-fludeoxyglucose (FDG) Positron Emission Tomography with Magnetic resonance imaging (PET/MRI) in participants with known metastatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Correlation of DWI and FDG to detect disease.

SECONDARY OBJECTIVE:

I. Inter-reader variability of DWI interpretation by region.

OUTLINE:

Participants will be imaged at a single timepoint using whole body DWI concurrent with FDG PET/MRI within 60 days of receiving a non-FDG PET (either PET/CT or PET/MRI). There will be an optional PET/MRI performed within six months of the original study. Participants will be followed up through a medical records review for up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Non FDG PET imaging study scheduled to be performed within 60 days (before or after) of the research PET/MRI.
3. Ability to understand a written informed consent document, and the willingness to sign it.
4. Diagnosis of metastatic cancer.

Exclusion Criteria:

1. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the Investigator to be unsuitable for participation.
2. Individuals with contraindications to MRI. This will be determined through review of the UCSF MRI screening form by qualified site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of lesions characterized as positive | Up to 6 months
  The overall proportion of lesions that will be characterized as positive on whole body (WB) diffusion weight imaging (DWI) and FDG PET.

SECONDARY OUTCOMES:
Inter-reader variability of diffusion weight imaging (DWI) interpretation | Up to 6 months
  Inter-reader variability is the degree of agreement among independent observers who rate, code, or assess the same image. Eighteen regions per participant will be scored by two blinded readers at each time point and assessed for the presence of DWI positive disease (local disease; nodal disease: pelvic, retroperitoneal, thoracic, and other; osseous disease: skull, ribs and sternum, cervical/thoracic/lumbar spine, right/left pelvis, sacrum and upper/lower extremities; visceral disease: lung, liver, and other). Scores range from 0 to 1 with 1 being excellent agreement between the two readers.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No